CLINICAL TRIAL: NCT05553886
Title: A Randomized, Double-blind, Positive-drug Parallel Controlled, Multicenter Phase III Trial of the Efficacy and Safety of S086 Tablets in Patients With Chronic Heart Failure With Reduced Ejection Fraction (HFrEF)
Brief Title: S086 Tablets for Chronic Heart Failure With Reduced Ejection Fraction
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Clinical study of S086 tablets
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, positive drug parallel control, multicenter
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S086 piece (Experimental): Sacubitril alisartan calcium tablets,60mg,120mg,180mg,240mg
  Interventions: Drug: To evaluate whether the efficacy of the study drug is noninferior to that of the positive control drug
- Sacubitril valsartan sodium tablets (Active Comparator): Sacubitril valsartan sodium tablets,50mg,100mg
  Interventions: Drug: To evaluate whether the efficacy of the study drug is noninferior to that of the positive control drug

INTERVENTIONS:
Drug: To evaluate whether the efficacy of the study drug is noninferior to that of the positive control drug — To evaluate whether the efficacy of the study drug is noninferior to that of the positive control drug

SUMMARY:
A randomized, double-blind, positive-drug parallel controlled, multicenter phase III trial of the efficacy and safety of S086 tablets in patients with chronic heart failure with reduced ejection fraction (HFrEF)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic heart failure (NYHA grade ⅱ-ⅳ) with reduced ejection fraction (LVEF≤40%) and elevated BNP were diagnosed 1a.
2. Patients received a stable dose of the underlying treatment for heart failure, defined as no change in dose for at least 4 weeks before screening 1b.
3. Volunteer to participate in the trial and sign an informed consent form 1c.

Exclusion Criteria:

1. Previous continuous administration of sacubitril valsartan sodium 150mg bid or more for more than 3 months 1a.
2. Use of other study drugs or use of any study medical device within 1 day of the visit or within 30 days prior to the visit or within 5 half-lives of the drug, whichever is longer 1b.
3. Known or suspected allergy to S086, sacubitril valsartan sodium, ARB, ACEI, or enkephin inhibitor (NEPI), and known or suspected contraindications to sacubitril valsartan sodium 1c.
4. A previous history of intolerance to the recommended target dose of ACEI or ARB 1d.
5. He had a history of angioedema 1e.
6. Acute coronary syndrome occurred within 6 weeks before visit 1 1f.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sacubitril valsartan sodium tablets (trade name: Nohintal) were used as a control to study the efficacy of S086 tablets in the treatment of Chronic heart failure with reduced ejection fraction（HFrEF）. | the end of 28th week
  Left ventricular ejection fraction (LVEF) changed from baseline at the end of 28th week,Normal result value 50-70%.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People' S Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No